CLINICAL TRIAL: NCT02669537
Title: Utility of the GoPro Hero 3 Camera as an Educational Tool For Vaginal Surgical Skills
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GoPro
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Hysterectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GOPRO resident (Experimental): Residents will use the gopro during a vaginal procedure, review the case with the attending after, and perform a 2nd case of the same type. The VVSI and GRS will be used to assess any changes in surgical skill
  Interventions: Device: GoPro Camera
- Control Resident (No Intervention): Residents will use standard surgical education practices, direct instruction from attending, surgical atlas, online videos. They will perform 2 cases of the same type and the difference in VVSI and GRS will be assessed
- GOPRO medical student (Experimental): Medical students will be allowed to watch the surgery on an iPad with the GoPro app. Their assessment of the educational value of the surgery will be assessed at the end of the procedure. They will also take a pre and post-test focusing on surgical instruments and steps used in the procedure.
  Interventions: Device: GoPro Camera
- Control Medical Student (No Intervention): Medical students will be taught using standard practices, i.e instruction by residents/attendings. Their assessment of the educational value of the surgery will be assessed at the end of the procedure. They will also take a pre and post-test focusing on surgical instruments and steps used in the procedure.

INTERVENTIONS:
Device: GoPro Camera — The gopro camera will be used to record the procedure which will be reviewed by the resident prior to performing a second procedure of the same type.
  Arms: GOPRO medical student; GOPRO resident

SUMMARY:
Utilization of the GoPro camera to facilitate vaginal surgical education among residents and medical students

DETAILED DESCRIPTION:
Surgical Skills Assessment:

Resident Control Group (Routine Educational Practice): Participants in this group will be exposed to routine surgical education as practiced at University Hospitals Case Medical Center, Department of OB/Gyn. This includes real time instruction at the time of surgery for the resident trainee performing all or part of the procedure as appropriate for their level of training. The resident may use any teaching tools before or after the surgery including online surgical videos, a surgical atlas or textbook. Immediately after the procedure the attending surgeon will evaluate the trainee using a validated 13-item Vaginal Surgical Skills Index (VSSI) form and the 7-item Global Rating Scale of Operative Performance (GRS) . The use of this scale is also part of standard surgical educational practice. The trainee will then perform an additional procedure of the same type within a 4 week period (the average duration of a rotation) and again undergo evaluation using the VSSI form by the attending surgeon. This is again part of routine educational practice in order to monitor progression of surgical skills.

Resident GoPro Group: Participants assigned this group will perform or assist with the procedure based on level of training and experience, as is usual practice in the residency training program. The resident surgeon will be wearing the camera (GoPro Hero 3) during the procedure. This is not part of routine practice. Immediately after the procedure the attending surgeon will evaluate the trainee using the VSSI and GRS forms. The trainee will then have a chance to review the video of their surgery with the attending surgeon within a 14-day period. The trainee will then perform a 2nd procedure of the same type within a 4 week period (the average duration of a rotation) and again undergo evaluation using the VSSI form by the attending surgeon. It is common for residents to perform a type of procedure (cerclage, culdoplasty, vaginal hysterectomy, etc.) many times during a rotation. However, for the purpose of the research study, we will only be comparing the change in the VVSI score between 2 procedures.

In both groups, surgical assistants will be instructed not to automatically assist but to wait for the participant to instruct them on what assistance they require.

The surgical skills inventory will be marked by the participant with their numerical designation and will then be placed in a locked box in the pre-operative area of the Humphrey operating room suite. These will be collected by the study investigators at the end of each week. The key to the box will be kept in a locked cabinet in Amy Schmidt's office on the 5th floor of MacDonald Women's Hospital.

Medical Student Evaluation of the OR Experience:

Medical students will be able to watch surgeries in real time using the GoPro App which will be downloaded to an iPad specifically purchased for use in this study. The video will be streamed over the secure UH BOYD network with both the surgeon and medical student are in the same operating room. The GoPro App does not allow the video to be saved to the iPAD.

At the end of each surgery medical student participants will be given a short survey with how satisfied they were with the level of teaching in the operating room (Appendix 3).

The survey will be marked by the participant with their numerical designation and will then be placed in a locked box in the pre-operative area of the Humphrey operating room suite. These will be collected by the study investigators at the end of each week. The key to the box will be kept in a locked cabinet in Amy Schmidt's office on the 5th floor of MacDonald Women's Hospital.

The results of the survey will be compared between those students viewing the surgery on the GoPro App and to those who are participating in the surgery without the GoPro camera. The survey is not routine educational practice, however, surveys are often employed in our department to gauge medical student attitudes.

Additionally all students who do not initially view a surgery with the GoPro app (those in the control group and those who choose not to participate in the research study) will be given the opportunity to use the GoPro app during a different surgery.

Acquisition of Surgical Video: Patients will be informed that the surgery will be recorded using a recording device and, if the patient chooses to allow recording, informed consent will be obtained using the standard image release consent form from UHCMC The video recording will not include any patient identifiers or markings.

ELIGIBILITY:
Inclusion Criteria:

* - Resident physician volunteers (PGY 1-4) currently in the OB/Gyn residency training program at University Hospitals Case Medical Center
* Medical student volunteers (MS1-MS4) currently enrolled at the Case Western Reserve University School of Medicine, Cleveland Clinic Lerner College of Medicine, or on an Ob/Gyn away rotation at the University Hospitals Case Medical Center

Exclusion Criteria:

* - Trainees who do not volunteer or do not wish to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in surgical skill score using the Vaginal Surgical Skills Inventory (VVSI) | 12 months
  Assessment of change in score between 2 consecutive procedures using the GoPro camera, compared to surgeons who did not use the camera
Change in score using the Global Rating Scale (GRS) | 12 months
  Assessment of change in score between 2 consecutive procedures using the GoPro camera, compared to surgeons who did not use the camera